CLINICAL TRIAL: NCT00254215
Title: The Effect of 4 Diets Varying in Glycemic Index, Glycemic Load, Carbohydrate and Protein, on Weight, Body Composition and Cardio-Vascular Risk Factors
Brief Title: Glycemic Load, Weight Loss and Cardiovascular Disease Risk
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Meat & Livestock Australia (Unknown); National Heart Foundation, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHF G02S 0768 - Brand-Miller
Record Dates: First submitted 2005-11-13; First posted 2005-11-15 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2005-07

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity; glycemic index; glycemic load; high protein diet; blood cholesterol
MeSH Terms: conditions — Overweight; Obesity

INTERVENTIONS:
Behavioral: high protein & low glycemic index diets

SUMMARY:
To investigate the hypothesis that reducing the glycemic load of the diet will improve changes in body composition and cardio-vascular risk factors. The study compares a conventional reduced-fat, high carbohydrate diet with 3 means of reducing glycemic load: changing the carbohydrates to low-GI choices, replacing some of the carbohydrate with protein, or combining both effects to produce the lowest glycemic load.

DETAILED DESCRIPTION:
Conventional low fat diets produce modest wegiht loss at best and the results are not well maintained. More recently there has been interest in low glycemic index and high protien diets wiht some evidence that these produce better fat loss and improvement in cardiovascular risk factors. This trial aims to evaluate these different approaches and compare the outcomes over 12 weeks. Major outcomes are weigth loss, body composition change, blood lipids change, measures of glucose homeostasis, insulin resistance, leptin and CRP.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age BMI >=25 stable weight for 3 months non-vegetarian good understanding of English

Exclusion Criteria:

medications other than the contraceptive pill weight >150kg (weight limit of DEXA machine) vegetarian (diets included red meat) specific diets diabetes or impaired glucose tolerance pregnancy

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120
Dates: Start 2002-03; Study Completion 2004-10

PRIMARY OUTCOMES:
weight loss at 12 weeks
Fat loss at 12 weeks
Lean mass change at 12 weeks

SECONDARY OUTCOMES:
Total cholesterol, LDL and HDL cholesterol change at 12 weeks
glucose, insulin & measures of insulin sensitivity change at 12 weeks
TG change at 12 weeks
Leptin change at 12 weeks
CRP change at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennie C Brand-Miller, PhD, Principal Investigator — University of Sydney
Locations (1):
- University of Sydney, Sydney, New South Wales, Australia

REFERENCES:
- [Result] McMillan-Price J, Petocz P, Atkinson F, O'neill K, Samman S, Steinbeck K, Caterson I, Brand-Miller J. Comparison of 4 diets of varying glycemic load on weight loss and cardiovascular risk reduction in overweight and obese young adults: a randomized controlled trial. Arch Intern Med. 2006 Jul 24;166(14):1466-75. doi: 10.1001/archinte.166.14.1466. PMID 16864756